CLINICAL TRIAL: NCT01401660
Title: Observational Study of the Electrophysiological Course of Low Back Pain Using CERSR® Imaging Technology
Brief Title: Study of Low Back Pain Using CERSR® Imaging Technology
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator withdrew from the study.
Sponsor: Verium Diagnostics, Inc. (Industry)
Responsible Party: Tamala J. Wampler / Vice President QA & RA, Verium Diagnostics, Inc.
Other Study IDs: SMI-2010-002; RP# 11002 (Other: Summa Health Systems IRB)
Record Dates: First submitted 2011-03-29; First posted 2011-07-25 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Low Back Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Subjects who do not currently have low back pain.
- Group B: Subjects who have low back pain at the time of the study, and who are currently being treated or have been previously treated for their low back pain and do not wish to receive further treatment for their pain.
- Group C: Subjects who have low back pain at the time of the study, and wish to receive physical therapy to reduce their low back pain.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The physician will complete a physical exam as well as analyze a completed CERSR® scan study to determine the root cause of the low back pain. The physician will then prescribe a targeted physical therapy regime to address the cause of the low back pain.
  Groups: Group C

SUMMARY:
The purpose of this research study is to measure with CERSR® (Computerized Electrophysiological Reconstruction of the Spinal Regions) the electrical signals made by the muscles in the lower back 1) when the subject has no low back pain 2) during the time low back pain begins, or 3) during the treatment and resolution of the low back pain, and 4) to study the changes which take place in these muscles as the pain improves with physical therapy treatment as an intervention. The hypotheses to be tested are 1) The CERSR® scan parameters for normal (pain-free) subjects are different from those of subjects with low back pain. 2) CERSR® scan aids the physician in determining a directed physical therapy treatment which leads to relief of low back pain following no more than eight weeks of physical therapy, as measured by relief of pain using a Visual Analog Scale and symptom improvement as measured using the Oswestry Disability Index.

DETAILED DESCRIPTION:
The purpose of this research study is to measure with CERSR® (Computerized Electrophysiological Reconstruction of the Spinal Regions) the electrical signals made by the muscles in the lower back 1) when the subject has no low back pain 2) during the time low back pain begins, or 3) during the treatment and resolution of the low back pain, and 4) to study the changes which take place in these muscles as the pain improves with physical therapy treatment as an intervention. The hypotheses to be tested are 1) The CERSR® scan parameters for normal (pain-free) subjects are different from those of subjects with low back pain. 2) CERSR® scan aids the physician in determining a directed physical therapy treatment which leads to relief of low back pain following no more than eight weeks of physical therapy, as measured by relief of pain using a Visual Analog Scale and symptom improvement as measured using the Oswestry Disability Index.

ELIGIBILITY:
Inclusion Criteria Groups A, B and C:

1. Male and female employees of the study center.
2. Between the ages of 18 and 70 years.
3. Current employees as well as new hires.

Exclusion Criteria Group A:

1. Low back pain.

Exclusion Criteria Group B:

1. Low back pain due to fracture, tumor, infection, cauda equina, severe neurological deficit.
2. Pregnant.
3. Sensitivity to isopropyl alcohol used to prepare the low back surface.
4. Inability to complete the required collection positions for the CERSR® scan.
5. Inability or unwillingness to adhere to the protocol and follow-up schedule.
6. Anyone under care of a physician for active liability or workman compensation cases.
7. Anyone who has had an open spinal procedure in the last three months.
8. Anyone who has undergone spine injections within the last two months.

Exclusion Criteria Group C:

1. Low back pain due to fracture, tumor, infection, cauda equina, severe neurological deficit
2. Pregnant.
3. Sensitivity to isopropyl alcohol used to prepare the low back surface.
4. Inability to complete the required collection positions for the CERSR scan.
5. Inability or unwillingness to adhere to the protocol and follow-up schedule.
6. Anyone under care of a physician for active liability or workman compensation cases.
7. Anyone who has had an open spinal procedure in the last three months.
8. Anyone who has undergone spine injections within the last two months.
9. Anyone who is currently undergoing physical therapy or chiropractic treatments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be selected from employees of Summa Health System. Current employees as well as new hires will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2011-05

PRIMARY OUTCOMES:
Change from Baseline in Pain Visual Analog Scale | Upon enrollment (day 1 - baseline) and four weeks and eight weeks
  The subjects will complete a form indicating their pain level upon enrollment. Subjects will then be scanned again at four weeks and at eight weeks. At the time of the scan subjects will also be asked to complete a follow up VAS. Upon completion of the study the change in VAS scores will be analyzed.

SECONDARY OUTCOMES:
Change from Baseline Oswestry Disability Index (ODI) | Upon enrollment (day 1 - baseline) and at four weeks and at eight weeks
  The subjects will complete the Oswestry Disability Index upon enrollment. Subjects will then be scanned again at four weeks and at eight weeks. At the time of the scan subjects will also be asked to complete a follow up ODI. Upon completion of the study the change in ODI scores will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Shah, M.D., Principal Investigator — Summa Health Systems
Locations (2):
- United States (2):
  - Summa Center for Clinical Trials, Akron, Ohio
  - Summa St. Thomas Hospital, Akron, Ohio

REFERENCES:
- [Background] Finneran MT, Mazanec D, Marsolais ME, Marsolais EB, Pease WS. Large-array surface electromyography in low back pain: a pilot study. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1447-54. doi: 10.1097/01.BRS.0000067565.16832.B9. PMID 12838104